CLINICAL TRIAL: NCT02707250
Title: Oblique Subcostal Transverses Abdominal Plane Block in Laparoscopic Cholecystectomy
Brief Title: Oblique Subcostal Tap Block Efficacy in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Breazu Caius Mihai, Dr.Breazu Caius Mihai MD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IuliuHatieganuU
Record Dates: First submitted 2016-02-19; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: pethidine; laparoscopic cholecystectomy; bupivacaine
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Oblique subcostal tap block with normal sterile saline ,20 ml, bilateral, single shot,24h
  Interventions: Drug: Placebo
- Bupivacaine (Active Comparator): Oblique subcostal tap block with bupivacaine 0,25% ,20 ml, bilateral, single shot,24h
  Interventions: Drug: Bupivacaine
- Pethidine (Active Comparator): Oblique subcostal tap block with pethidine 1% ,10 ml,bilateral,single shot,24h
  Interventions: Drug: Pethidine
- Pethidine Local Infiltration (L.I.) (Active Comparator): Local infiltration of pethidine 1% at trocar insertion sites, 5ml /site, 24h compared with Tap Block with pethidine 1%
  Interventions: Drug: Pethidine Local Infiltration (L.I)

INTERVENTIONS:
Drug: Placebo — Tap Block performed with normal sterile saline 20 ml on the right side and 20 ml on the left side
  Other Names: Tap Block Placebo
  Arms: Placebo
Drug: Bupivacaine — Tap Block performed with Bupivacaine 0,25% 20 ml on the right side and 20 ml on the left side.
  Other Names: Tap Block Bupivacaine
  Arms: Bupivacaine
Drug: Pethidine — Tap Block performed with pethidine 1% 10 ml on the right side and 10 ml on the left side
  Other Names: Tap Block Pethidine
  Arms: Pethidine
Drug: Pethidine Local Infiltration (L.I) — Local infiltration of port sites (trocar insertion sites) with pethidine 1% 5ml each port (trocar site) ,4 ports total 20 ml pethidine 1%
  Other Names: Pethidine Local Infiltration
  Arms: Pethidine Local Infiltration (L.I.)

SUMMARY:
Laparoscopic cholecystectomy although a minimally invasive procedure, may be accompanied by considerable pain after surgery. More recently transversus abdominis plane (TAP) block was extensively studied as a potential analgesic maneuver after laparoscopic cholecystectomy. The subcostal approach (OSTAP block) is a variation on the TAP block that produces reliable supraumbilical analgesia.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is a minimally invasive widespread surgical procedure, with postoperative lower pain scores and quick recovery of the patient. However some of patients may complain of considerable pain after surgery . There are several approaches to postoperative pain management after laparoscopic cholecystectomy such as patient-controlled analgesia with opioids (IV-PCA), neuraxial blocks, intraperitoneal injection of local anesthetics, wound infiltration, each being more or less effective, with specific side effects.

The transversus abdominis plane block (TAP-Block) is a regional analgesia technique that comes as an alternative to "classical" procedures of postoperative analgesia. Described by Rafi and McDonnell et al. this technique has undergone some changes over times, which increased its efficiency. Thus, Hebbard et al. described ultrasound subcostal oblique approach (OSTAP) of the block allowing analgesia in both the upper and lower abdomen, with a lower rate of complications due to the direct ultrasound visualization. Different studies confirmed the analgesic efficacy of this technique and the postoperative opioid sparing effect after laparoscopic cholecystectomy .

Traditionally, the transversus abdominis plane block is achieved with classical amino-amides local anesthetics, bupivacaine, levobupivacaine and ropivacaine being the most commonly used .

Based on the local anesthetic properties of pethidine, a synthetic opioid, our study aimed to evaluate prospectively the analgesic efficacy of pethidine in achieving transversus abdominis plane block by ultrasound oblique subcostal approach in patients scheduled for elective laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) I-II
* Age over 18years old
* patients scheduled elective laparoscopic cholecystectomy

Exclusion Criteria:

* Open cholecystectomy - excluded due to increased levels of pain in open procedures
* Renal dysfunction (Serum Cr > 1.2) - excluded due to potential altered metabolism of anesthetic and pain medications
* Coagulopathy or anticoagulation - increased risk of bleeding from nerve block injection
* Allergy or contraindication to any of the study medications or anesthetic agents
* Chronic opioid analgesic use at home - excluded due to potential difficulty in assessing pain caused by the procedure alone
* Patient inability to properly describe postoperative pain to investigators (language barrier, dementia, delirium, psychiatric disorder)
* Pregnancy
* Prisoners
* Patient or surgeon refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | Recorded 2 hours postoperative
  This outcome is measured with a visual analogue scale (VAS, from 0 to 10) at 2 hours postoperative, while the patient is in his bed. This outcome is recorded in and compared between all four groups.
Pain Scores | Recorded 6 hours postoperative
  This outcome is measured with a visual analogue scale (VAS, from 0 to 10) at 6 hours postoperative, while the patient is in his bed. This outcome is recorded in and compared between all four groups.
Pain Scores | Recorded 12 hours postoperative
  This outcome is measured with a visual analogue scale (VAS, from 0 to 10) at 12 hours postoperative, while the patient is in his bed. This outcome is recorded in and compared between all four groups.
Pain Scores | Recorded 24 hours postoperative
  This outcome is measured with a visual analogue scale (VAS, from 0 to 10) at 24 hours postoperative, while the patient is in his bed. This outcome is recorded in and compared between all four groups.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | 0-4 hours
  Recording total amount of intraoperative fentanyl consumption
Time to first opioid administration in Post Anesthetic Care Unit | 0-4 hours postoperative
  Recording time to first opioid administration in post aesthetic care unit
Cumulative opioid consumption | Recorded in the first 24 hours perioperative period
  Recording total amount of opioids used in postoperative period
Side effects | Recorded in the first 24 hours postoperative
  nausea, vomiting, pruritus and sedation on a 4 point scale as none, mild, moderate and severe

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ionescu, MD, Study Director — University of Medicine and Pharmacy "Iuliu Hatieganu" Cluj-Napoca,Romania
Locations (1):
- Regional Institute of Gastroenterology and Hepatology "Prof.dr.Octavian Fodor", Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Breazu C, Margarit S, Bartos A, Ionescu D. Postoperative Analgesia after Laparoscopic Cholecystectomy - Prospective, Randomized, Double Blind, Control Trial. Chirurgia (Bucur). 2022 Oct;117(5):563-571. doi: 10.21614/chirurgia.2769. PMID 36318686